CLINICAL TRIAL: NCT07151170
Title: Telerehabilitation Versus Supervised Pelvic Floor Muscle Training in Postmenopausal Women With Urinary Incontinence
Brief Title: Telerehabilitation Versus Supervised Pelvic Floor Muscle Training in Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aliza Tahir
Record Dates: First submitted 2025-08-24; First posted 2025-09-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Urinary Incontinence; Urinary Incontinence,Stress; Urinary Incontinence, Urge; Postmenopausal Symptoms
Keywords: Pelvic Floor Muscle Training; Telerehabilitation; Supervised Exercise; Postmenopausal Women; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: There will be comparison between the two groups, experimental and control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Pelvic Floor Muscle Taining (TR-PFMT) Group (Experimental): This group will receive a 6-week standardized Pelvic Floor Muscle Training program (18 sessions, 2/week, 60 min) delivered online by a physiotherapist. The program includes patient education on pelvic floor anatomy, bladder habits, and lifestyle advice, along with diaphragmatic breathing, pelvic mobility, and progressive strengthening of phasic and tonic Pelvic Floor Muscle fibers in multiple positions. Home exercises are prescribed with gradual progression, and participants submit weekly exercise diaries for monitoring and motivation.
  Interventions: Other: Telerehabilitation Pelvic Floor Muscle Training (TR-PFMT) Group
- Supervised Pelvic Floor Muscle Training (S-PFMT) Group (Active Comparator): In the supervised group, the protocol will be delivered by a physiotherapist in a clinical environment by face-to-face. The same standardized Pelvic Floor Muscle Training protocol will be monitored exactly the same as TR-PFMT.
  Interventions: Other: Supervised Pelvic Floor Muscle Training (S-PFMT) Group

INTERVENTIONS:
Other: Telerehabilitation Pelvic Floor Muscle Training (TR-PFMT) Group — The program will be delivered online in small groups by a physiotherapist. The program includes diaphragmatic breathing, pelvic mobility (pelvic tilts, hip circles, cat-cow), stretching (butterfly, child pose, deep squat), and progressive strengthening of phasic and tonic fibers through stationary PFMT (10-sec moderate-hold + 3 quick flicks, 8 sets in weeks 1-3, 10 sets in weeks 4-6, 10-sec rest) and home-based PFMT (10 fast contractions and 10 moderate-hold contractions, 2 sets in weeks 1-2 with weekly set increases, 10-sec rest), performed in prone lying, supine hook-lying, butterfly, sitting, and standing positions. All sessions will be recorded, and participants will submit weekly exercise diaries.
  Arms: Telerehabilitation Pelvic Floor Muscle Taining (TR-PFMT) Group
Other: Supervised Pelvic Floor Muscle Training (S-PFMT) Group — In the supervised group, the protocol will be delivered by a physiotherapist in a clinical environment by face-to-face. The standardized Pelvic Floor Muscle Training protocol will be monitored exactly the same as Telerehabilitation group (TR-PFMT).
  Arms: Supervised Pelvic Floor Muscle Training (S-PFMT) Group

SUMMARY:
Urinary Incontinence (UI) is a prevalent condition impacting women across all age groups, varing in both severity and type. Urinary Incontinence affects 25%-45% of women worldwide. A systematic review explains that menopause-driven estrogen decline leads to atrophy of pelvic floor muscles (PFM). The goal of this randomized controlled trial is to compare the effects of telerehabilitation-based pelvic floor muscle training with a supervised face-to-face pelvic floor muscle training program in improving urinary incontinence symptoms, pelvic floor muscle funtion and quality of life (QoL) in postmenopausal women. Participnts will be randomly assigned to one of the two groups, and both will receive an identical standardized pelvic floor muscle training protocol. The results of this clinical trial will help evaluate how telerehabilitation can provide support for postmenopausal women with urinary incontinence and improve health outcomes.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is common among postmenopausal women and is characterized by involuntary urine leakage, leading to physical, psychological, and social challenges. Its prevalence increases after menopause due to hormonal changes, along with loss of connective tissue and muscle fiber degradation. This results in reduced maximal voluntary contraction and diminished coordination, contributing to increased UI risk in postmenopausal women. Postmenopausal women with UI present significantly increased pelvic floor muscle (PFM) stiffness both at rest and during contraction, signalling structural deterioration. Therefore this increased stiffness, linked to tissue atrophy, compromises muscle contraction and is closely associated with reduced urethral support. Systematic reviews highlight that postmenopausal women often are marginalized or grouped with wider age ranges, limiting the significance of outcomes to this specific demographic. Therefore adequately powered randomized controlled trails directly comparing Tele-rehabilitation and supervised Pelvic floor muscle training (PFMT) in postmenopausal women are limited. PFMT is the first-line conservative treatment recommended by international guidelines. Traditionally, PFMT is delivered in supervised, in-person sessions with a physiotherapist; however, hurdles such as mobility issues, transportation costs can reduce access to supervised sessions. Tele-rehabilitation may overcome these barriers by offering flexible and home-based treatment. Tele-rehabilitation, using secure video conferencing to deliver PFMT in real time, may improve accessibility, adherence, and convenience. Hence evaluating the effectiveness and acceptability of remote PFMT in postmenopausal women is both timely and clinically important. This study will provide stronger statistical power to address the existing evidence gap and contribute to the growing field of digital physiotherapy by providing valuable evidence evaluating whether Tele-rehabilitation can serve as an effective and feasible alternative to face-to-face intervention for managing urinary incontinence in postmenopausal women, thereby improving women's health outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women between the ages of 45-65.
* Postmenopausal status, defined as absence of menstruation for more than 12 months.
* Experiencing symptomatic urinary incontinence, indicated by a Questionnaire for Urinary Incontinence Diagnosis (QUID) score greater than "0".
* Able to comprehend and accurately respond to the questionnaire (i.e., no language barriers) and reading and writing Urdu language.
* Free from any physical or psychological conditions that could hinder participation in the study.
* Participants must have access to both the internet and a mobile phone/laptop
* Signing the informed consent form.

Exclusion Criteria:

* Women with cognitive impairments, neurological disorders, pelvic malignancies.
* Individuals with a history of intra-abdominal and pelvic surgery or radiation therapy.
* Presence of active urinary tract/vaginal infection
* Presence of incontinence except stress and urge urinary incontinence (e.g. overflow incontinence or dribbling urine after urination)
* Presence of voiding dysfunction (e.g. incomplete voiding, intermittent urination or delay in starting to urinate)
* Women with contraindications to pelvic floor muscle training (e.g., pelvic pain resulting from endometriosis, coccydynia or anismus, unexplained vaginal bleeding and anal fissure).
* Women aged over 65 years
* Body mass index ≥ 27.4 kg/m²
* Currently undergoing hormone therapy
* Lack of pelvic floor muscle contraction ability (pelvic floor muscle strength <2 according to the Modified Oxford Scale)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) score | Baseline and 6 weeks
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a valid, widely used tool to assess urinary incontinence (UI) symptoms, severity and its impact on quality of life. It has three scored items (leakage frequency, amount, and interference) and one unscored diagnostic item identifying possible causes or situations of leakage (e.g., coughing, sneezing, exertion). Scores range from 0-21, with higher scores showing greater severity: slight (1-5), moderate (6-12), severe (13-18), very severe (19-21)
Change in pelvic floor muscle strength using the Modified Oxford Scale | Baseline and 6 weeks
  The Modified Oxford Scale is a validated grading system used to assess pelvic floor muscle strength through vaginal palpation. It ranges from 0 to 5. The Modified Oxford Scale developed by Laycock is scored as, a score of 0: indicates no contraction, 1: a slight flicker, 2: a weak squeeze, 3: a moderate contraction with some lift, 4: a good contraction with resistance, and 5: a strong contraction with firm resistance and lift. Higher grades indicate stronger pelvic floor muscles.
Change in Urinary Impact Questionnaire short form (UIQ-7) score | Baseline and 6 weeks
  The Urinary Impact Questionnaire short form (UIQ-7) is a validated self-report tool. The UIQ-7 consists of 7 items assessing how urinary incontinence affects daily activities, emotional health, and social interactions. Each item is scored from 0 (not at all) to 3 (greatly), giving a total score of 0-21, with higher scores indicating greater negative impact.
Change in Incontinence Impact Questionnaire, Short Form (IIQ-7) score | Baseline and 6 weeks
  The IIQ-7 emphasises the functional impact of incontinence, comprising 7 items that evaluate the influence of incontinence on physical activity, travel, social relationships, and emotional health. Each response is scored 0-3, resulting in a total score of 0-21, where higher scores indicate a more severe impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Principal Investigator — Riphah International University, Islamabad, Pakistan
Locations (2):
- Pakistan (2):
  - Riphah International Hospital, Islamabad, Islamabad
  - Pakistan Railway Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Berre M, Filiatrault J, Reichetzer B, Dumoulin C. Group-Based Pelvic Floor Telerehabilitation to Treat Urinary Incontinence in Older Women: A Feasibility Study. Int J Environ Res Public Health. 2023 May 11;20(10):5791. doi: 10.3390/ijerph20105791. PMID 37239520
- [Background] Lin KY, Chen CY, Wu PC, Huang MH, Ou YC, Kao YL, Lin KH. The feasibility and effects of a telehealth-delivered physical therapy program for postmenopausal women with urinary incontinence: A pilot mixed-methods study. Maturitas. 2025 Jun;197:108376. doi: 10.1016/j.maturitas.2025.108376. Epub 2025 Apr 23. PMID 40286562
- [Background] Parra NS, Jaramillo AP, Zambrano J, Segovia D, Castells J, Revilla JC. The Effectiveness of Pelvic Floor Muscle Exercise in Urinary Incontinence: A Systematic Literature Review and Meta-Analysis. Cureus. 2023 Sep 11;15(9):e45011. doi: 10.7759/cureus.45011. eCollection 2023 Sep. PMID 37720131